CLINICAL TRIAL: NCT01788904
Title: Plasma i-FABP as Predictor for Irreversible Bowel Ischemia After Interventional Re-vascularization in Patients With Acute Mesenteric Ischemia
Brief Title: Plasma i-FABP as Predictor for Irreversible Bowel Ischemia
Acronym: FARAMIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Regensburg (Other)
Collaborators: William Cook Europe (Industry)
Responsible Party: Principal Investigator, Peter Heiss, Peter Heiss, MD, MS, University Hospital Regensburg
Other Study IDs: FARAMIS 2013
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Acute Mesenteric Ischemia; Bowel Necrosis
Keywords: Acute mesenteric ischemia; Percutaneous endovascular revascularization; Intestinal plasma fatty acid binding protein (i-FABP); Bowel necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma, blood serum, EDTA blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute mesenteric ischemia: Patients with acute mesenteric ischemia meeting the in-/exclusion criteria

SUMMARY:
In the FARAMIS study, we aim to investigate the longitudinal course of intestinal plasma fatty acid binding protein (i-FABP) in patients with acute mesenteric ischemia (AMI) undergoing primary percutaneous angiographic intervention.

The investigators postulate that patients with fully re-established intestinal blood flow and vital intestines will display a significant drop of plasmatic i-FABP within 24 hours, while patients requiring subsequent intestinal resection due to irreversible bowel necrosis will not.

If true, patients requiring laparotomy and bowel resection could be identified and patients in whom angiographic intervention led to successful cure of disease would not be exposed to potentially perilous surgery.

DETAILED DESCRIPTION:
Intestinal plasma fatty acid binding proteins (i-FABP) have been introduced as a powerful marker for the diagnosis of intestinal ischemia. Based on several small studies, this marker is referred to as a sensitive indicator for intestinal ischemia. I-FABP is characterized by its short half-time of eleven minutes in blood circulation, which might allow "real-time" monitoring of necrotic intestinal segments.

Subjects meeting the in-/exclusion criteria will undergo five to six blood collections: one baseline assessment before revascularization, three assessments directly after angiographic intervention (5/30/120 minutes), and one assessment after 24 hours. An additional blood collection will be performed in patients who underwent subsequent surgery. In addition, clinical exams of the patient are carried out.

Subjects will be observed for 72 hours after percutaneous revascularization and retrospectively classified depending on the clinical course: recovering patients or patients undergoing surgery without signs of necrotic segments will be attributed to group A. Patients in whom intestinal necrosis is confirmed by surgery or autopsy will belong to group B. For all patients, clinical and laboratory findings will be reported in a descriptive manner.

To evaluate whether the post-interventional course of plasmatic i-FABP is a reliable predictor for successful revascularization, the minimum level of i-FABP at the time points 5, 30 and 120 Minutes is divided by the baseline (= before intervention) level of i-FABP. This ratio (R) reflects the decrease (or increase) of i-FABP after revascularization. Receiver operating characteristic (ROC)-analysis will be carried out and the area under the curve will be determined for different R-values (e.g. 0.3, 0.5, 0.7).

We postulate that patients with fully re-established intestinal blood flow and vital intestines will display a significant drop of plasmatic i-FAPB within 24 hours, while patients requiring subsequent intestinal resection due to irreversible bowel necrosis will not.

ELIGIBILITY:
Inclusion Criteria:

* Presence of acute mesenteric ischemia due to stenosis of the superior mesenteric artery, thromboembolization of the superior mesenteric artery, non-occlusive mesenteric ischemia or acute portal vein thrombosis (as confirmed by CT scan)
* The vascular anatomy is suitable for percutaneous revascularization
* A primary endovascular re-vascularisation approach is intended based on an interdisciplinary decision by the visceral surgeon, the vascular surgeon and interventional radiologist. This therapeutic decision is made independently of the proposed FARAMIS study.
* A peripheral or central line is present to perform repeated blood collections

Exclusion Criteria:

* Clinically or imaging results indicating that perforation of the bowel is present or suspected
* Hemodynamic instability (shock)
* Pre-existing severe liver or kidney damage (defined as spontaneous international normalized ratio >2 or creatinine >2 mg/dl.)
* Anemia with hemoglobin concentration < 7g/dl
* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Post-interventional course of plasmatic i-FABP as reliable predictor for successful bowel revascularization | 72 hours
  Subjects will be observed for 72 hours after percutaneous revascularization. Patients will then be divided into two groups: patients not requiring surgery and not dying from intestinal necrosis will be allocated to group A. Subjects who undergo surgery without signs of necrotic segments will also be attributed to group A. Patients in whom intestinal necrosis is confirmed by surgery or autopsy will belong to group B.
  To evaluate whether the post-interventional course of plasmatic i-FABP is a reliable predictor for successful revascularization, the minimum level of i-FABP at the time points 5, 30 and 120 Minutes is divided by the baseline (= before intervention) level of i-FABP. This ratio (R) reflects the decrease (or increase) of i-FABP after revascularization. ROC-analysis will be carried out and the area under the curve will be determined for different R-values.

SECONDARY OUTCOMES:
Baseline level of i-FABP as predictor of bowel necrosis | 72 hours

OTHER OUTCOMES:
Levels of i-FABP, interleukine 6 and 8 | 72 hours
  Association of increased levels of i-FABP, interleukine 6 and 8 with extension of intestinal necrosis according to the pathology report and occurrence of organ failure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Heiss, MD, MS, Principal Investigator — University Hospital Regensburg Germany
Locations (1):
- University Hospital Regensburg, Regensburg, Germany